CLINICAL TRIAL: NCT04794517
Title: Evaluating the Short-term Renal and Systemic Effects of Dapagliflozin in Non-diabetic Patients With Stage IV CKD at Risk of ESKD Because of Severe Renal Insufficiency and Persistent Proteinuria
Brief Title: Dapagliflozin in Non-diabetic Stage IV CKD
Acronym: ADAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ADAPT; 2021-000726-10 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney disease; Proteinuria; Dapagliflozin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMP (Experimental): Dapagliflozin 10 mg/die will be administered orally for six-weeks.
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Placebo (Placebo Comparator): Placebo, one tablet/die will be administered orally for six-weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Dapagliflozin 10 mg/die will be administered orally for six-weeks.
  Arms: IMP
Other: Placebo — Placebo one tablet/die will be administered orally for six-weeks.
  Arms: Placebo

SUMMARY:
This is a phase 2b, prospective, randomized, cross-over, double-blind, placebo-controlled trial primarily aimed at assessing whether the SGLT2 inhibitor dapagliflozin ameliorates hyperfiltration and reduces proteinuria as compared to placebo in patients with non-diabetic CKD, with particular focus on those at highest risk of progression to end stage kidney disease (ESKD) because of severe renal insufficiency (Stage IV CKD) and proteinuria (>0.5 g/24 hours). The study will also evaluate renal and systemic mechanisms mediating treatment effects on GFR and will explore biochemical factors possibly mediating these effects.

DETAILED DESCRIPTION:
As chronic kidney disease (CKD) continues to increase worldwide, along with the demand for related life-saving therapies, the financial burden of CKD will place an increasing drain on health care systems. Experimental studies showed that glomerular capillary hypertension and impaired sieving function with consequent protein overload play a pathogenic role in the progression of CKD. Consistently, human studies show that proteinuria is an independent predictor of progression and that its reduction is renoprotective. At comparable BP control, inhibitors of the renin-angiotensin system (RAS), including angiotensin converting enzyme (ACE) inhibitors and angiotensin II receptor blockers (ARBs), more effectively than non-RAS inhibitor therapy reduce proteinuria, slow progression to ESRD, and even improve the kidney function achieving disease regression in some cases. In participants with diabetes, RAS inhibitors delay the onset of microalbuminuria and its progression to macroalbuminuria, and ACE inhibitors may reduce the excess cardiovascular mortality associated with diabetic renal disease. In addition to RAS inhibitors, however, multimodal approaches including lifestyle modifications and multidrug therapy will be required in most cases to optimize control of the several risk factors for CKD and related cardiovascular morbidity. Novel medications, including proximal tubular sodium - glucose co-transporter -2 (SGLT2 inhibitors - that ameliorate glomerular hyperfiltration and proteinuria and slow renal disease progression in type 2 diabetes by mechanisms apparently independent of improved metabolic control - might help further improve the cost-effectiveness of renoprotective interventions even in non-diabetic CKD. This phase 2, prospective, randomized, cross over, placebo-controlled trial will primarily aim to assess whether the SGLT2 inhibitor dapagliflozin ameliorates hyperfiltration and reduces proteinuria as compared to placebo in patients with non-diabetic CKD, with particular focus on those at highest risk of progression to end stage kidney disease (ESKD) because of severe renal insufficiency (Stage IV CKD) and proteinuria (>0.5 g/24 hours).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female more than 18 year old
3. Non-diabetic Stage-IV CKD
4. Fasting blood glucose ≤ 125 mg (≤ 6.9 mmol/l) and HbA1C ≤6.4% (≤ 47 mmol/mol)58 without treatment with oral blood glucose lowering medications and/or insulin
5. Two-hour plasma glucose <200 mg/dl during 75-g oral glucose tolerance test (OGTT)58
6. Persistent proteinuria (24-hour urinary protein excretion ≥ 0.5 grams in at least two consecutive evaluations >1 week apart) despite RAS inhibitor therapy with ACE inhibitors and/or ARBs (or without RAS inhibitors in patients with specific contraindications to these medications)
7. eGFR 15 to 30 ml/min/1.73 m2 by CKD-Epi equation
8. Blood pressure <150/90 mmHg without changes in blood pressure lowering medications over the last four weeks before the randomization
9. Negative pregnancy test (urine or serum) for female subjects of childbearing potential.10
10. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of dapagliflozin\placebo to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.
11. Male subjects must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of IMP to prevent pregnancy in a partner.
12. Subjects who are blood donors should not donate blood during the study and for 3 months following their last dose of dapagliflozin\placebo.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Participation in another clinical study with an investigational product during the last month
3. Ischemic kidney disease (because of possible excess risk of acute kidney injury upon SGLT2-inhibitor associated reduction in sodium pool and kidney perfusion pressure)
4. Rapidly progressive kidney disease (e GFR reduction ≥ 30% over the last three months) and expected risk of progression to end stage kidney failure and need of renal replacement therapy by dialysis or transplantation during the study period.
5. Active systemic autoimmune diseases;
6. Concomitant treatment with steroids or any other immunosuppressive agent
7. Hypersensitivity to the active principle (dapagliflozin) or any of the excipients (e.g. lactose);
8. Severe/unstable heart failure with or without decreased systolic function requiring hospitalization or changes in pharmacological therapy over the last three months
9. Uncontrolled hypertension (BP >150/90 mmHg despite optimized pharmacological treatment and diet or symptomatic hypotension
10. Positive hepatitis C antibody hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening
11. Known to have tested positive for human immunodeficiency virus
12. Drug or alcohol abuse
13. Inability to fully understand the possible risks and benefits related to study participation
14. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 90 days after last dose; or intending to donate ova during such time period;
15. If male, the subject intends to donate sperm while on the study this study or for 90 days after last dose;
16. Participation in another interventional clinical trial within the 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration rate (GFR) | Changes from baseline and day 1, 8, 42,84, 92,126 and 140.
  GFR measured by the Iohexol plasma clearance technique
24-hour urinary protein excretion | Changes from start (day 0, day 84) and end (day 42, day 126) of each Treatment Period with dapagliflozin or placebo
  24-hour urinary protein excretion will be measured as median of three measurements in three consecutive 24-hour urine collections

SECONDARY OUTCOMES:
Renal plasma flow (RPF) | Changes from baseline and day 1, 8, 42,84, 92,126 and 140.
  RPF will be assessed by the Para Amino Hippuric (PAH) plasma clearance technique.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No